CLINICAL TRIAL: NCT01553266
Title: Mobile Diabetes Education Teams in Primary Care
Status: Completed | Type: Observational
Sponsor: Toronto Metropolitan University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Trillium Health Centre (Other)
Responsible Party: Principal Investigator, Enza Gucciardi, Assistant Professor, Toronto Metropolitan University
Other Study IDs: REB 2010-282; 247888 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2012-02-29; First posted 2012-03-14 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2013-12

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus; diabetes care; diabetes self-management education; primary care physicians; interprofessional collaboration; diabetes education programs; qualitative; quantitative; implementation; evaluation; health services; coordinated care; integrated care; patient care processes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- MDET intervention
  Interventions: Behavioral: Mobile Diabetes Education Teams intervention
- Control group: Patients who have not received the MDET intervention.

INTERVENTIONS:
Behavioral: Mobile Diabetes Education Teams intervention — A MDET (one Registered Nurse and Registered Dietician) supports primary care physicians by providing diabetes management education to the PCPs' patients onsite, one to four times a month based on patient volume.
  Other Names: MDET
  Groups: MDET intervention

SUMMARY:
The purpose of this study is to evaluate the implementation of the Mobile Diabetes Education Team (MDET) intervention in the Greater Toronto Area, as well as the intervention's effectiveness in improving patient clinical and care process outcomes.

The study's hypotheses are that the MDET intervention results in the following outcomes:

* Improvement in patient clinical outcomes;
* An increase in the proportion of primary care physicians (PCPs) performing patient care processes according to clinical practice guidelines;
* An increase in the proportion of referrals to, and patients' utilization of, diabetes education programs (DEPs).

DETAILED DESCRIPTION:
The proposed research is the first evaluation of the implementation of Mobile Diabetes Education Teams (MDETs) in Canada. This intervention will support primary care providers (PCPs) by offering a diabetes education team (one registered nurse [RN] and one registered dietitian [RD]) one to four times a month, based on patient volume, at various primary care sites to assist in and share the care and management of patients with diabetes. This intervention is in collaboration with the Mississauga Halton Local Health Integration Network (MH LHIN) and will be hosted by Trillium Diabetes Management Centre and Halton Diabetes Program. Each hosting site received permanent operational funding for half a diabetes education team (salary support) from the Ontario Ministry of Health and Long-term Care (MHLTC) under the new Ontario Diabetes Strategy.

The rationale for incorporating MDETs in primary care was guided by the extensive literature on the underuse and low referral to diabetes education programs (DEPs), where diabetes self-management education is primarily offered. Low utilization is due to low PCP referral rates to these services, as well as numerous systematic and operational barriers for both PCPs and patients. Consequently, the majority of Canadians are receiving diabetes care solely from their PCPs, who have expressed barriers to caring for diabetes patients and are providing sub-optimal care as they are not consistently adhering to clinical practice guidelines. As a result, MHLTC is investing millions of dollars in expanding and aligning current programs to increase access to team-based care.

The objective of this research is to evaluate a structural redesign in how the investigators deliver diabetes care and self-management education using a collaborative approach between PCPs and DEPs guided by the Chronic Care Model as a conceptual framework. The purpose of this research is twofold: 1) to evaluate the effects of MDET intervention on: (i) patient clinical outcomes; (ii) quality of care patients receive from PCPs; (iii) PCPs' referral to and their patients' utilization of DEPs; and 2) to assess the implementation processes of the MDET intervention and the degree of collaboration and team functioning between PCPs and the MDET members across primary care sites. A mixed-methods approach is proposed over a three year period.

Patients will be referred to the MDET by PCPs. The MDET will meet with patients for two hours (one hour with the RN and one hour with the RD) to assess the level of diabetes knowledge, diabetes self-care and lifestyle habits; this data will be used to develop patient treatment priorities and action care plans. Three 30 minute follow-up visits with the MDET will be carried out over a one-year period for all patients where patient action plans are reviewed, discussed and potentially revised. A communication tool has been developed to better facilitate communication of patient information between PCPs and MDETs. Case conferences will be conducted when major changes are to be made to the patient's treatment plan after a patient's visit. Accordingly, PCPs and educators are collaboratively managing patient care.

A cluster-randomized trial stepped wedge design will be used to ensure all sites will eventually receive the intervention, while still facilitating the comparison of change within individuals and between study groups across time points that is attributed to the intervention. The inclusion criteria for reviewing patient medical records are patients who are over 18 years of age, have type 2 diabetes, and have an HbA1c of greater than 8%. Twenty unique patient chart extractions will be performed at 0, 6, 12, 18, 24 months from 12 primary care sites to collect patient care processes and patient clinical outcome data (for a total of 1,200 patient charts). Characteristics of interprofessional collaboration between PCPs and the MDET will be assessed at each practice site at the end of one year. To assess the implementation of the MDET across sites, qualitative process data, such as in-depth interviews with patients, PCPs and the MDETs, and MDETs' field notes and debriefing sessions will be analyzed.

MDETs will strengthen and formalize links between primary care providers and diabetes education programs within the community, increase patient access to diabetes self-management education and support, and potentially improve patient experience and clinical outcomes through enhanced coordination and integration of care. This study is timely and relevant as DEPs and local PCPs are starting to integrate services across Canada; thus, our research will provide the evidence necessary to inform practice of such a model. If results are promising, this model can be extended to direct how those with impaired glucose tolerance and gestational diabetes/post-gestational diabetes; and as a result, diabetes prevention, management and care are delivered, and can greatly reduce the burden of diabetes in Canada.

ELIGIBILITY:
Inclusion Criteria:

* Has Diabetes Mellitus, Type 2;
* Is 18 years of age or older;
* Has an HbA1c of > 8%.

Exclusion Criteria:

* Has type of diabetes that requires intense and specialized treatment, such as Type 1 diabetes, gestational diabetes, or patients on a multiple, daily insulin regime.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Those living with diabetes
Sampling Method: Non-Probability Sample
Enrollment: 900 (Actual)
Dates: Start 2012-03-01 (Actual); Primary Completion 2014-03-12 (Actual); Study Completion 2017-04-12 (Actual)

PRIMARY OUTCOMES:
Change from 12 months prior to intervention in HbA1c up to 12 months during the intervention | At 12 months prior to intervention; up to 12 months during the intervention
  Change in patients' results for HbA1c from 12 months prior to intervention up to 12 months during the intervention.

SECONDARY OUTCOMES:
Change from 12 months prior to intervention in low-density lipoprotein (LDL-C) up to 12 months during the intervention | At 12 months prior to intervention; up to 12 months during the intervention
  Change in patients' results for low-density lipoprotein (LDL-C) from 12 months prior to intervention up to 12 months during the intervention.
Change from 12 months prior to intervention in total cholesterol-high density lipoprotein ratio (TC-HDL ratio) up to 12 months during the intervention | At 12 months prior to intervention; up to 12 months during the intervention
  Change in patients' results for total cholesterol-high density lipoprotein ratio (TC-HDL ratio) from 12 months prior to intervention up to 12 months during the intervention.
Change from 12 months prior to intervention in blood pressure up to 12 months during the intervention | At 12 months prior to intervention; up to 12 months during the intervention
  Change in patients' results for blood pressure from 12 months prior to intervention up to 12 months during the intervention.
Change from 12 months prior to intervention in testing for HbA1c up to 12 months during the intervention | At 12 months prior to intervention; up to 12 months during the intervention
  Change in proportion of primary care physicians testing for patients' HbA1c from 12 months prior to intervention up to 12 months during the intervention.
Change from 12 months prior to intervention in blood pressure testing up to 12 months during the intervention | At 12 months prior to intervention; up to 12 months during the intervention
  Change in proportion of primary care physicians testing for patients' blood pressure from 12 months prior to intervention up to 12 months during the intervention.
Change from 12 months prior to intervention in lipid profile testing up to 12 months during the intervention | At 12 months prior to intervention; up to 12 months during the intervention
  Change in proportion of primary care physicians testing for patients' lipid profile from 12 months prior to intervention up to 12 months during the intervention.
Change from 12 months prior to intervention in nephropathy screening up to 12 months during the intervention | At 12 months prior to intervention; up to 12 months during the intervention
  Change in proportion of primary care physicians screening patients for nephropathy (ACR and eGFR) from 12 months prior to intervention up to 12 months during the intervention.
Change from 12 months prior to intervention in foot exams up to 12 months during the intervention | At 12 months prior to intervention; up to 12 months during the intervention
  Change in proportion of primary care physicians performing foot exams from 12 months prior to intervention up to 12 months during the intervention.
Change from 12 months prior to intervention in dilated retinal exam referrals up to 12 months during the intervention | At 12 months prior to intervention; up to 12 months during the intervention
  Change in proportion of primary care physicians referring patients to dilated retinal exams from 12 months prior to intervention up to 12 months during the intervention.
Change from 12 months prior to intervention in flu vaccine provision or recommendation up to 12 months during the intervention | At 12 months prior to intervention; up to 12 months during the intervention
  Change in proportion of primary care physicians providing for, or recommending, the flu vaccine to patients from 12 months prior to intervention up to 12 months during the intervention.
Change from 12 months prior to intervention in Diabetes Education Program referrals at 12 months of intervention | 12 months prior to intervention to 12 months of the intervention
  Change in primary care physicians' referrals to, and patients' utilization of, diabetes education programs from 12 months prior to the intervention at 12 months of the intervention.
Patient attendance at scheduled MDET visits | At 12 months of intervention
  Number of MDET appointments planned for each patient compared to the number of MDET visits attended.
Collaborative Practice Assessment Tool scores of PCPs and MDET educators in intervention | At 12 months of intervention
  Collaborative Practice Assessment Tool scores of PCPs and MDET educators at 12 months of the intervention, to assess interprofessional collaboration between PCPs and educators.
Patients' interview responses regarding intervention effectiveness | At 12 months of intervention
  In-depth interview responses of 20 randomly-selected patients at 12 months of the intervention, regarding the usefulness of the intervention in better understanding their condition, diabetes self-management strategies, and convenience and quality of delivery.
PCPs' interview responses regarding interprofessional collaboration in, and the implementation of, the intervention | At 12 months of intervention
  In-depth interview responses of 16 randomly-selected PCPs at 12 months of the intervention, regarding their experiences with the intervention, their collaboration and teamwork, barriers and facilitators to implementation, and suggestions to improve the intervention.
MDET educators' interview responses regarding interprofessional collaboration in, and the implementation of, the intervention | At 12 months of intervention
  In-depth interview responses of 16 randomly-selected educators at 12 months of the intervention, regarding their experiences with the intervention, their collaboration and teamwork, barriers and facilitators to implementation, and suggestions to improve the intervention.
MDET educators' reflective journal responses regarding interprofessional collaboration in, and the implementation of, the intervention | Up to 2 years
  MDET educators' monthly field notes in their reflective journals regarding their experiences and reflections of those experiences with the implementation of, and interprofessional collaboration in, the intervention.
MDET educators' quarterly debriefing session group discussions regarding intervention issues | Up to 2 years
  MDET educators' group discussions during MDET debriefing sessions, held quarterly, regarding any issues with the implementation of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Enza Gucciardi, PhD, Principal Investigator — Toronto Metropolitan University

REFERENCES:
- [Derived] Gucciardi E, Fortugno M, Horodezny S, Lou W, Sidani S, Espin S, Webster F, Shah BR. Will Mobile Diabetes Education Teams (MDETs) in primary care improve patient care processes and health outcomes? Study protocol for a randomized controlled trial. Trials. 2012 Sep 13;13:165. doi: 10.1186/1745-6215-13-165. PMID 22974080